CLINICAL TRIAL: NCT03047837
Title: A Randomized, Phase II, Double-blind, Placebo-controlled, Multicenter, 2x2 Factorial Design Biomarker Tertiary Prevention Trial of Low-dose Aspirin and Metformin in Stage I-III Colorectal Cancer Patients. the ASAMET Trial
Brief Title: A Randomized, 2x2 Factorial Design Biomarker Prevention Trial of Low-dose ASA and Metformin in Stage I-III Crc Patients
Acronym: ASAMET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of enrolment
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Responsible Party: Principal Investigator, Andrea DeCensi, Principal Investigator, Ente Ospedaliero Ospedali Galliera
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 27UCS2015; 2015-004824-77 (EudraCT Number)
Record Dates: First submitted 2017-02-01; First posted 2017-02-09 (Estimated); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Tertiary Prevention in Colon Cancer
Keywords: Colorectal cancer; aspirin; metformin; chemoprevention
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): placebo Aspirin (1 tablet daily) + placebo Metformin (1 tablet BID) for 12 months
  Interventions: Other: Placebo
- Metformin (Experimental): placebo Aspirin (1 tablet daily) + active Metformin (850 mg, 1 tablet BID), for 12 months
  Interventions: Drug: MET
- Aspirin (Experimental): active Aspirin (100 mg, 1 tablet daily) + placebo Metformin (1 tablet BID), for 12 months
  Interventions: Drug: ASA
- Apirin plus Metformin (Experimental): active Asprin (100 mg, 1 tablet daily) + active Metformin (850 mg, 1 tablet BID), for 12 months
  Interventions: Drug: ASA; Drug: MET

INTERVENTIONS:
Drug: ASA — Arm C (experimental arm) Treatment: active ASA + placebo MET Dose: 100 mg, 1 tablet daily + 1 tablet twice a day (BID) Duration: 12 months
  Other Names: Cardioaspirin
  Arms: Apirin plus Metformin; Aspirin
Drug: MET — Arm B (experimental arm) Treatment: placebo ASA + active MET Dose: 1 tablet daily+ 850 mg, 1 tablet twice a day (BID) Duration: 12 months
  Other Names: Metformin
  Arms: Apirin plus Metformin; Metformin
Other: Placebo — Arm A (control arm) Treatment: placebo ASA + placebo MET Doses: 1 tablet daily +1 tablet twice a day (BID) Duration: 12 months
  Arms: Placebo

SUMMARY:
It has been shown that Aspirin (ASA) as well as Metformin (Met) can inhibit the incidence and mortality of colorectal cancer (CRC). In this randomized, placebo controlled clinical trial we compare the effect of these two drugs alone and their combination to prevent recurrent CRC after surgery.

DETAILED DESCRIPTION:
Epidemiological studies and cardiovascular prevention trials have shown that low-dose aspirin (ASA) can inhibit colorectal cancer (CRC) incidence and mortality, including inhibition of distant metastases. Metformin (MET) has also been associated with decreased CRC incidence and mortality in meta-analyses of epidemiological studies in diabetics and has been shown to decrease by 40% colorectal adenoma recurrence in a randomized trial. Recent studies have shown that ASA is an inhibitor of mTOR/S6K1 and an activator of AMPK, targeting regulators of intracellular energy homeostasis and metabolism, and that the combination of ASA and MET, another AMPK activator and S6K1 inhibitor, has a striking additive effect on AMPK activation and mTOR inhibition, with increased autophagy and decreased cell growth in CRC cell lines. While both drugs are being tested as single agents, their combination has not been tested in trials.

This is a randomized, placebo-controlled, double blind, 2x2 biomarker trial of ASA and MET to test the activity of either agent alone and the potential synergism of their combination on a set of surrogate biomarkers of colorectal carcinogenesis. After surgery 160 patients with stage I-III colon cancer will randomly be assigned in a four-arm trial to either ASA, 100 mg day, MET 850 mg bid, their combination, or placebo for one year. The primary endpoint biomarker is the change, defined as the difference between pre- and post-treatment expression of nuclear factor kappa-B (NFκB), in the unaffected mucosa of proximal and distal colon obtained by multiple biopsies in two paired colonoscopies one year apart. Additional biomarkers will include: 1) the genomic profile of candidate genes, pathways, and overall genomic patterns in tissue biopsies by genome wide gene expression arrays; 2) the IHC expression of tissue pS6K, p53, beta-catenin, PI3K; 3) the associations of mutations and SNPs with treatment response by next generation sequencing of primary tumors; 4) the measurement of circulating IL-6, CRP and VEGF and 5) plasma and colonic MET concentrations and their correlation with biomarker profiles.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 and ≤ 80 years.
* Patients with completely resected stage I, II, or III primary colorectal cancer within 24 months prior to randomization, regardless of (neo-)adjuvant chemotherapy. Patients with pT1 CRC treated with endoscopic polypectomy.
* Adjuvant chemotherapy and (neo-)adjuvant radiotherapy terminated at least 3 months before randomization.
* ECOG performance status ≤ 1.
* Satisfactory hematological and biochemical functions:

  * Platelets ≥ 100 x 10^9/L
  * Creatinine clearance estimated with the Cockcroft - Gault formula ≥ 60 mL/min. Patients with Gault formula ≥ 45-59 ≤ ml/min are eligible but they will receive a single (evening) tablet of MET, 850 mg.
  * AST and ALT ≤ 2.5 times ULN.
* Females of childbearing potential/males with partners of childbearing potential participating in the study are to use effective methods of birth control during study participation. Female participants must provide a pregnancy test, according to local/national guidelines.
* Able to understand and sign an informed consent (or have a legal representative who is able and willing to do so).

Exclusion Criteria:

* Patients who are not able to undergo colonoscopy.
* Patients who are allergic or intolerant to ibuprofen or naproxen,or who have MET-, or ASA-, or salicylate intolerance or more generalized drug intolerance to non-steroidal anti-inflammatory drugs (NSAIDs).
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing or participating in the study and/or comply with study procedures.
* Chronic treatment with ASA or other NSAIDs or MET or patients who are on current long term treatment (≥ 4 consecutive weeks) with ASA, NSAID or COX -2 inhibitors or MET.
* Diabetic patients on drug treatment are excluded.
* Anticoagulant therapy (dicumarol, heparin, fondaparinux, apixaban, dabigatran etexilate, rivaroxaban) or active current treatment with antiplatelet agents (e.g. off-study ASA, clopidogrel, prasugrel, ticagrelor, or ticlopidine).
* Any other invasive malignancies (with the exclusion of basal cell carcinoma or cutaneous squamous cell carcinoma) diagnosed during the last 5 years before randomization. Past history of any other invasive CRC than the one the patient is currently being treated for
* Alcohol or drug abuse.
* Prior history of gastro-intestinal bleeding or hemorrhagic diathesis (e.g. hemophilia).
* Erosive-ulcerative lesions in the gastrointestinal tract.
* History of erosive GERD or active erosive GERD on gastroscopy.
* Concomitant corticosteroid treatment.
* Known deficiency of glucose-6-phosphate dehydrogenase (G6PD).
* Treatment with another investigational drug < 28 days prior to study entry.
* Concurrent participation in a clinical trial with the same endpoints.
* History of hemorrhagic stroke.
* Lynch Syndrome (HNPCC).
* Crohn's disease (CD) and Ulcerative Colitis (UC).
* Pregnant or lactating females.
* History of lactic acidosis.
* Liver dysfunction including chronic active hepatitis and cirrhosis not compensated.
* History of vitamin B12 deficiency or megaloblastic anemia.
* Uncontrolled coronary syndrome or symptomatic congestive heart failure (e.g. Class III or IV New York Heart Association's Functional Classification).
* Inability or unwillingness to swallow tablets.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
NFκB | 1 year
  It will be measured the change, defined as the difference between post- and pre-treatment levels, in NFκB expression in normal colonic tissue. The NFκB transcription factor family is composed of the p65, RelB, c-Rel, p105, andt p100 subunits, and activation of the NFκB pathway is defined by the nuclear translocation of the p65 subunit. Therefore, cytoplasmic and nuclear localization of p65 will be immunohistochemically assessed as an indicator of NFκB activity. The analysis of expression will be performed by semi quantitative assessment: NFκB expression will be measured primarily as the percentage of positive nuclear areas for NFkB over the total nuclear areas in 10 section fields.

SECONDARY OUTCOMES:
pS6K, p53, beta-catenin, PI3K | 1 year
  It will be measured the change (defined as above) in IHC expression levels of pS6K, p53, beta-catenin, PI3K (from colon unaffected biopsy specimen). These biomarkers will be measured as described above for NFκB.
IL-6, CRP, VEGF and HOMA index | 1 year
  The change in circulating biomarkers IL-6, CRP, VEGF and HOMA index[homeostasis model assessment (fasting blood glucose (mmol/L)*insulin (mU/L))/22.5] will be measured in plasma and serum at two time points, pre- and post-intervention, using monoclonal ELISA kits.
Gene expression levels | 1 year
  Gene expression levels of candidate genes and pathways, in normal colonic tissue, will be measured on a genome-wide basis using Illumina HumanHT-12 Expression BeadChips targeting more than 47,000 transcripts including known splice variants across the human transcriptome.
Metformin concentration | 1 Year
  The blood and tissue MET levels will be measured. LC-MS/MS system will be used for the drug level determinations to be correlated with biomarker modulation and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Censi, MD, Principal Investigator — E.O. Ospedali Galliera
Locations (1):
- Medical Oncology Ente Ospedaliero Ospedali Galliera, Genova, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petrera M, Paleari L, Clavarezza M, Puntoni M, Caviglia S, Briata IM, Oppezzi M, Mislej EM, Stabuc B, Gnant M, Bachleitner-Hofmann T, Roth W, Scherer D, Haefeli WE, Ulrich CM, DeCensi A. The ASAMET trial: a randomized, phase II, double-blind, placebo-controlled, multicenter, 2 x 2 factorial biomarker study of tertiary prevention with low-dose aspirin and metformin in stage I-III colorectal cancer patients. BMC Cancer. 2018 Dec 4;18(1):1210. doi: 10.1186/s12885-018-5126-7. PMID 30514262